CLINICAL TRIAL: NCT02720991
Title: A Pilot Study of the Acceptability and Feasibility of an Out-patient Regimen of Medical Abortion With Mifepristone and 400 mcg Sublingual Misoprostol at 71-77 and 78-84 Days Gestation
Brief Title: A Pilot of an Outpatient Regimen of Medical Abortion With Mifepristone and Sublingual Misoprostol in the 11 and 12 Weeks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Hopital La Rabta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1014
Record Dates: First submitted 2016-03-10; First posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Abortion, 3 Months
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mifepristone and sublingual misoprostol (Experimental): 200 mg mifepristone and 400 ug sublingual misoprostol
  Interventions: Drug: Mifepristone; Drug: Sublingual misoprostol

INTERVENTIONS:
Drug: Mifepristone — 200 mg of oral mifepristone
  Other Names: miropristone; Mifeprex; Mifegyn
Drug: Sublingual misoprostol — 400 ug of misoprostol sublingually following mifepristone
  Other Names: cytotec

SUMMARY:
A pilot study on the acceptability and feasibility with Mifepristone and 400 mg of sub-lingual Misoprostol between 71-77 and 78-84 days of gestation for 50 cases.

DETAILED DESCRIPTION:
The study will enroll 25 women in each gestational age group. All participants will be submitted to routine screening as per current practice at La Rabta Hospital. The eligible women will receive a dose of 200 mg of mifepristone and 400 ug of misoprostol to take at home sublingually .

The first 5 women enrolled in each gestational age group will be asked to return to the clinic 24-48 hours after the initial visit to take misoprostol at the clinic and wait during a 3 hour observational period before returning to their homes. After this initial phase, the women will be asked to self-administer the misoprostol at home 24-48 hours after the administration of mifepristone and to return to the clinic 7-10 days later. At follow-up, a healthcare provider will assure her that her medical abortion is complete and after will ask women to respond to a series of questions in an exit interview.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 71-84 days of amenorrhea
* Seeking abortion services
* Prepared and able to sign the consent forms
* Accept to conform to study procedures and scheduled visits

Exclusion Criteria:

* Does not meet study criteria

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Acceptability of an ambulatory medical abortion treatment of 200 mg of mifepristone orally followed b 400 mcg of sublingual misoprostol at home, based on responses to questionnaire | 1 week

SECONDARY OUTCOMES:
Level of tolerance of side effects, based on responses to questionnaire | 1 week

IPD SHARING:
Plan to Share IPD: No